CLINICAL TRIAL: NCT06868745
Title: Randomized Clinical Trial: Effects of Melatonin Supplementation on Sleep Quality in Patients With Advanced Glaucoma
Brief Title: Effects of Melatonin Supplementation on Sleep Quality in Patients With Advanced Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Priscilla Fernandes Nogueira, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 36946620.9.0000.5505
Record Dates: First submitted 2025-01-25; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Glaucoma; Sleep Disturbance; Circadian Rhythm; Melatonin; Actigraphy
Keywords: glaucoma; sleep disturbance; circadian rhythm; melatonin; actigraph
MeSH Terms: conditions — Glaucoma; Parasomnias

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, parallel, cross-over, and double-blind therapeutic-type clinical study was conducted at the Glaucoma Division and the Department of Psychobiology at the Federal University of São Paulo - UNIFESP/EPM and the Eye Hospital Visao Laser in Santos/SP. The study involved 64 patients, with an age range of over 40 and under 80 years old. All participants underwent a complete ophthalmological evaluation and completed questionnaires on sleep quality (PSQI-BR), the Epworth Sleepiness Scale, and the Vision Function Questionnaire (NEI VFQ-25). Each participant received either 5mg of melatonin or a placebo for 30 days at different times. During this period, they were assessed using actigraphy, questionnaires, and examinations on day 0 (before starting the medication) and on day 30. Afterward, the use of the medication was discontinued.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: there is no
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- melatonin treatment group (Experimental): Each participant received melatonin 5 mg and placebo for a period of 30 days
  Interventions: Drug: Experimental: melatonin treatment group; Drug: Placebo comparator: placebo treatment group
- placebo treatment group (Placebo Comparator): Each participant received melatonin 5 mg and placebo for a period of 30 days
  Interventions: Drug: Experimental: melatonin treatment group; Drug: Placebo comparator: placebo treatment group

INTERVENTIONS:
Drug: Experimental: melatonin treatment group — Each participant received melatonin 5 mg for a period of 30 days
Drug: Placebo comparator: placebo treatment group — Each participant received placebo for a period of 30 days

SUMMARY:
A prospective, randomized, parallel, crossover, double-blind therapeutic clinical trial was conducted in accordance with the principles of the Resolution nº 466/12 of the National Health Council and was approved by the Ethics and Research Committee of the Federal University of São Paulo, project CEP/UNIFESP n:1023/2020, CAAE: 36946620.9.0000.5505. Written informed consent was obtained from all participants. The study was conducted at the Glaucoma Division and the Department of Psychobiology at the Federal University of São Paulo - UNIFESP/EPM and at the Laser Vision Eye Hospital - Santos/SP between May/2022 and July/2023.

DETAILED DESCRIPTION:
The study included 64 patients with a diagnosis of advanced primary open-angle glaucoma in both eyes.

Patients were classified as glaucoma cases if they had at least 3 repeatable, consecutive, abnormal visual field test results, defined as a pattern standard deviation (PSD) outside the 95% normal confidence limits or a Glaucoma Hemifield Test (GHT) result outside normal limits matching the appearance of the optic disc, presenting a Mean deviation of <-12.00 dB in the better eye(7,14,17), according to the Hoddap-Parish-Anderson classification for glaucoma severity, using the SITA-Standard strategy, with no involvement of the fixation region (absence of statistically significant points in the central 5º for both total and pattern deviation).

Patients were considered as glaucomatous if they had signs of glaucomatous optic neuropathy based on optic disc stereophotographs. Evidence of glaucomatous damage to the optic disc nerve was considered if they had RNFL defects or localized or diffuse neuroretinal rim loss. There were 32 participants in the melatonin group and 32 in the placebo group. The age range of the volunteers was over 40 years and under 80 years.

Subjects were excluded if they were younger than 40 or older than 80 years; best-corrected visual acuity of less than 0.4 logMAR; Patients who work at night or recently traveled across time zones, use topical or systemic medications that could disrupt circadian rhythms, for example Benzodiazepines, Non-benzodiazepines (hypnotics), Sedative antidepressants, Melatonin and melatonin agonists, patients with previously defined obstructive sleep apnea or other disorders such as depression and insomnia were excluded. Only patients with an open angle on gonioscopy were included in our study.

Each participant received melatonin 5 mg and placebo for a period of 30 days at different time points. The packages were identical, each labeled with the letters F and I. Only the supervisor Dr. Augusto Paranhos Junior, had knowledge of which package contained the original drug. Additionally, the pills within the packages were identical and supplied by the same researcher, who was not informed about the significance of the letters on the packaging.

On day 0 (D0 - before starting the medication), subjects completed the Pittsburgh Sleep Quality Index (PSQI) and the Epworth Sleepiness Scale (ESS) to assess subjective sleep quality and daytime sleepiness, respectively. At D0, they also completed the 25-Item National Eye Institute Visual Function Questionnaire (NEI VFQ-25). The 24-hour daily profile of sleep parameters was assessed on a single night by actigraphy.

Questionnaires and actigraphy assessments were carried out, 30 days after each medication and in the wash out interval 7 days discontinuing the use of the medication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Primary Open-Angle Glaucoma: Must have a confirmed diagnosis of primary open-angle glaucoma.
* Cup-to-Disc Ratio > 0.6: The ratio of cup to disc on optic disc imaging must be greater than 0.6.
* Visual Acuity ≥ 0.4 logMAR: Participants must have a visual acuity of 0.4 logMAR or better in the better eye.
* Age: Participants must be aged 40 to 80 years, inclusive.

Exclusion Criteria:

* Pregnancy: Female participants who are pregnant or planning to become pregnant during the study period.
* Current or Past Diagnosis of Depression: Participants with a current or past history of depression.
* Corneal or Retinal Diseases: History or active disease of the cornea or retina (e.g., diabetic retinopathy, macular degeneration).
* Shift Work: Participants who work night shifts or irregular hours.
* Travel Across Time Zones: Participants who have traveled across time zones in the last 30 days prior to enrollment.
* Diagnosed Obstructive Sleep Apnea: History of obstructive sleep apnea or a current diagnosis of the condition.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Effects of Melatonin Replacement on Sleep Quality of Patients with Advanced Glaucoma | From enrollment to the end of treatment in 2 months
  To compare the quality of sleep in patients with advanced glaucoma after 30 days of melatonin 5 mg and 30 days of placebo. The comparison of efficacy between groups will be assessed based on the improvement in sleep quality between medications.

SECONDARY OUTCOMES:
Effects of Melatonin Replacement on Sleep Quality of Patients with Advanced Glaucoma | From registration to the end of treatment in 2 months
  To compare the effects on sleep quality after using melatonin 5 mg and placebo. The effects on sleep quality will be measured by the following assessments: questionnaire (Pittsburgh Sleep Quality Index). Sleep quality is measured on a 7-level scale, with the last level being the worst rating;
Effects of Melatonin Replacement on Sleep Quality of Patients with Advanced Glaucoma | From registration to the end of treatment in 2 months
  To compare the quality of sleep in patients with advanced glaucoma after 30 days of melatonin 5 mg and 30 days of placebo. The comparison of efficacy between groups will be assessed based on the improvement in sleep quality between medications, using the actigraph, which will analyze the total sleep time through minutes slept, between the groups, the longer the time slept, the better quality of sleep, and also analyzes the number of awakenings, how many times during sleep the patient wakes up, the greater the number of awakenings, the worse the quality of sleep.
Effects of Melatonin Replacement on Sleep Quality of Patients with Advanced Glaucoma | From registration to the end of treatment in 2 months
  To compare the effects on sleep quality after using melatonin 5 mg and placebo. The effects on sleep quality will be measured by the following assessments: questionnaire, Epworth Sleepiness Scale, level of excessive sleepiness is measured on 8 levels, with the last level being the worst rating;
Effects of Melatonin Replacement on Sleep Quality of Patients with Advanced Glaucoma | From registration to the end of treatment in 2 months
  To compare the effects on sleep quality after using melatonin 5 mg and placebo. The effects on sleep quality will be measured by the following assessments: questionnaire, 25-Item National Eye Institute Visual Function Questionnaire, quality of life is measured on 25 levels, with the last level being the best rating.

CONTACTS AND LOCATIONS:
Locations (1):
- Casa, Santos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the publication of the results
Supporting Information: Study Protocol, ICF
Time Frame: concluded
Access Criteria: Word file by email